CLINICAL TRIAL: NCT00777088
Title: Pipeline for Uncoilable or Failed Aneurysms
Acronym: PUFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVPUFS0398
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Intracranial Aneurysm
Keywords: neurovascular embolization; therapeutic embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pipeline (Experimental): Placement of Pipeline Embolization Device in the parent artery at the aneurysm location
  Interventions: Device: Pipeline Embolization Device (PED)

INTERVENTIONS:
Device: Pipeline Embolization Device (PED) — 1 or more PEDs placed in the parent artery of the affected aneurysm via endovascular approach

SUMMARY:
To determine the safety and effectiveness of Pipeline Embolization Device for the treatment of uncoilable or failed wide-necked intracranial aneurysms (IA).

DETAILED DESCRIPTION:
Patients with large or giant aneurysms of the internal carotid artery treated with PED. Angiographic follow-up occurs at 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years, inclusive
* Patient has a single target IA in the anterior or posterior circulation that:

  a) Is located in the following regions of the internal carotid artery: i. Paraophthalmic (including paraclinoid, ophthalmic and hypophyseal segments) ii. Cavernous iii. Petrous

  b) Has a neck >4 mm or no discernible neck AND a size (maximum fundus diameter) >10 mm

  c) Has a parent vessel with diameter 2.5 - 5.0 mm distal/proximal to the target IA
* Subject has provided written informed consent using the Institutional Review Board (IRB)-approved consent form
* Subject has the necessary mental capacity to participate and is willing and able to comply with protocol requirements

Exclusion Criteria:

* More than one IA requires treatment in the next 6 months
* Subarachnoid hemorrhage from target IA in the past 60 days
* Unstable neurologic deficit (i.e., any worsening of clinical condition in the last 30 days)
* Irreversible bleeding disorder
* Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
* Inability to tolerate, documented evidence of adverse reaction or contraindication to study medications
* Stent in place at the target IA
* Contraindication to CT scan or MRI
* Allergy to contrast used in angiography that cannot be medically controlled
* Known severe allergy to platinum or cobalt/chromium alloys
* Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
* Woman of child-bearing potential who cannot provide a negative pregnancy test
* Evidence of active infection at the time of treatment
* Other conditions of the heart, blood, brain or intracranial vessels that carry a high risk of neurologic events (e.g., severe heart failure, atrial fibrillation, known carotid stenosis)
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments to 180 days
* Extracranial stenosis greater than 50% in the carotid artery for anterior circulation aneurysms
* Intracranial stenosis greater than 50% in the treated vessel

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2014-09-22 (Actual); Study Completion 2014-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Bescke, MD, Principal Investigator — New York University
Locations (10):
- United States (8):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Rush University, Chicago, Illinois
  - Central Du Page Hospital, Winfield, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - New York University, New York, New York
  - Stony Brook University, Stony Brook, New York
- National Institute of Neurosurgery, Budapest, Hungary
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Becske T, Potts MB, Shapiro M, Kallmes DF, Brinjikji W, Saatci I, McDougall CG, Szikora I, Lanzino G, Moran CJ, Woo HH, Lopes DK, Berez AL, Cher DJ, Siddiqui AH, Levy EI, Albuquerque FC, Fiorella DJ, Berentei Z, Marosfoi M, Cekirge SH, Nelson PK. Pipeline for uncoilable or failed aneurysms: 3-year follow-up results. J Neurosurg. 2017 Jul;127(1):81-88. doi: 10.3171/2015.6.JNS15311. Epub 2016 Oct 14. PMID 27739944
- [Derived] Sahlein DH, Fouladvand M, Becske T, Saatci I, McDougall CG, Szikora I, Lanzino G, Moran CJ, Woo HH, Lopes DK, Berez AL, Cher DJ, Siddiqui AH, Levy EI, Albuquerque FC, Fiorella DJ, Berentei Z, Marosfoi M, Cekirge SH, Kallmes DF, Nelson PK. Neuroophthalmological outcomes associated with use of the Pipeline Embolization Device: analysis of the PUFS trial results. J Neurosurg. 2015 Oct;123(4):897-905. doi: 10.3171/2014.12.JNS141777. Epub 2015 Jul 10. PMID 26162031

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pipeline
Started | 108
Completed | 107
Not Completed | 1
Not completed — PED Treatment not attempted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pipeline
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 18
  Hungary | 14
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Occurrence of Major Ipsilateral Stroke or Neurologic Death and Occurrence of Ipsilateral Stroke or Neurologic Death.
Description: The number of participants with occurrence of major ipsilateral stroke or neurologic death after PED placement at 180-days and the occurrence of ipsilateral stroke or neurologic death after Pipeline Embolization Devices (PED) placement at 5-years.
Time Frame: 180-days and 5-years
Population: Patients treated with one or more Pipeline Embolization Devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline
Number analyzed (Participants) | 107
Participants
  180-Days | 6
  5-Years | 10
Statistical Analysis 1: Comparison: Pipeline; Test type: Non-Inferiority — The cumulative rate of ipsilateral stroke or neurologic death is not ≥ 20% at 180-day clinical follow-up and the cumulative rate of ipsilateral stroke or neurovascular death is not ≥ 25% at 5-year clinical follow-up; p < .001, Bayesian

2. Primary Outcome: Count of Intracranial Aneurysms (IA) Evaluated as Completely Occluded (100%) Without Major Parent Artery Stenosis.
Description: The count of Intracranial Aneurysms (IA) evaluated as completely occluded (defined as Raymond Grade 1) without major parent artery stenosis at 180 days. The Raymond-Roy Grade scale measures the amount of visual contrast flow throughout the aneurysm anatomy. The Raymond-Roy aneurysm occlusion scale is follows:
  Complete = complete occlusion, no flow of contrast seen in the sac Residual Neck = partial occlusion, some flow, or eddying flow, in the sac Residual Aneurysm = incomplete occlusion, apparent flow into the sac
Time Frame: 180 days
Population: A total of 104 participants and 106 intracranial aneurysms treated with the Pipeline Embolization Device were included in the primary effectiveness endpoint analysis.
Measure: Count of Units; unit: Fully Occluded Intracranial Aneurysms
Units Other Than Participants: Fully Occluded Intracranial Aneurysms
Arm/Group | Pipeline
Number analyzed (Participants) | 104
Number analyzed (Fully Occluded Intracranial Aneurysms) | 106
Fully Occluded Intracranial Aneurysms | 78
Statistical Analysis 1: Comparison: Pipeline; Test type: Non-Inferiority or Equivalence — The rate of complete IA occlusion without major parent artery stenosis exceeds 50% with a posterior probability >0.975; p < 0.001, Bayesian

3. Secondary Outcome: Count of Intracranial Aneurysms (IA) Evaluated as Completely Occluded (100%) at 1 Year
Description: The count of Intracranial Aneurysms (IA) Evaluated as Completely Occluded (100%) (defined as Raymond-Roy grade 1) 1 year follow-up visit. The Raymond-Roy Grade scale measures the amount of visual contrast flow throughout the aneurysm anatomy. The Raymond-Roy aneurysm occlusion scale is follows:
  Complete = complete occlusion, no flow of contrast seen in the sac Residual Neck = partial occlusion, some flow, or eddying flow, in the sac Residual Aneurysm = incomplete occlusion, apparent flow into the sac
Time Frame: 1 Year
Population: Pipeline treated subjects with observable data at 1 year
Measure: Count of Units; unit: Target Intracranial Aneurysms
Units Other Than Participants: Target Intracranial Aneurysms
Arm/Group | Pipeline
Number analyzed (Participants) | 91
Number analyzed (Target Intracranial Aneurysms) | 91
Target Intracranial Aneurysms | 79

4. Secondary Outcome: Count of Intracranial Aneurysms (IA) Evaluated as Completely Occluded (100%) at 3 Year Follow-up
Description: The count of Intracranial Aneurysms (IA) evaluated as completely occluded (100%) (defined as Raymond-Roy grade 1) at 3 year follow-up. The Raymond-Roy Grade scale measures the amount of visual contrast flow throughout the aneurysm anatomy. The Raymond-Roy aneurysm occlusion scale is follows:
  Complete = complete occlusion, no flow of contrast seen in the sac Residual Neck = partial occlusion, some flow, or eddying flow, in the sac Residual Aneurysm = incomplete occlusion, apparent flow into the sac
Time Frame: 3 years
Population: Pipeline treated Subjects with observable data at 3 years
Measure: Count of Units; unit: Target Intracranial Aneurysms
Units Other Than Participants: Target Intracranial Aneurysms
Groups:
- Pipeline: Placement of Pipeline Embolization Device in the parent artery at the aneurysm location Pipeline Embolization Device (PED): 1 or more PEDs placed in the parent artery of the affected aneurysm via endovascular approach
Arm/Group | Pipeline
Number analyzed (Participants) | 76
Number analyzed (Target Intracranial Aneurysms) | 76
Target Intracranial Aneurysms | 71

5. Secondary Outcome: Count of Intracranial Aneurysms (IA) Evaluated as Completely Occluded (100%) at 5 Years
Description: The count of Intracranial Aneurysms (IA) evaluated as completely occluded (100%) (defined as Raymond-Roy grade 1) at 5-year follow-up. The Raymond-Roy Grade scale measures the amount of visual contrast flow throughout the aneurysm anatomy. The Raymond-Roy aneurysm occlusion scale is follows:
  Complete = complete occlusion, no flow of contrast seen in the sac Residual Neck = partial occlusion, some flow, or eddying flow, in the sac Residual Aneurysm = incomplete occlusion, apparent flow into the sac
Time Frame: 5 years
Population: Pipeline treated subjects with observable data at 5 years
Measure: Count of Units; unit: Target Intracranial Aneurysms
Units Other Than Participants: Target Intracranial Aneurysms
Arm/Group | Pipeline
Number analyzed (Participants) | 62
Number analyzed (Target Intracranial Aneurysms) | 62
Target Intracranial Aneurysms | 59

6. Secondary Outcome: Stenosis of the Parent Artery in PED at 3 Years
Description: Parent artery stenosis (narrowing of the artery from which the aneurysm arises) at 3-year follow-up
Time Frame: 3-years
Population: Subjects that completed imaging at the 3-year follow-up were included in the parent artery stenosis analysis.
Measure: Count of Units; unit: Parent Artery Assessments
Units Other Than Participants: Parent Artery Assessments
Arm/Group | Pipeline
Number analyzed (Participants) | 85
Number analyzed (Parent Artery Assessments) | 85
Parent Artery Assessments
  Stenosis 0 - 25% | 67
  Stenosis > 25 - 50% | 8
  Stenosis >50% - 75% | 0
  Stenosis >75% | 3
  Indeterminate | 7

7. Secondary Outcome: Stenosis of the Parent Artery in PED at 5 Years
Description: Parent artery stenosis at 5-year follow-up
Time Frame: 5-years
Population: Subjects that completed imaging at the 5-year follow-up were included in the parent artery stenosis analysis.
Measure: Count of Units; unit: Parent Artery Assessments
Units Other Than Participants: Parent Artery Assessments
Arm/Group | Pipeline
Number analyzed (Participants) | 64
Number analyzed (Parent Artery Assessments) | 64
Parent Artery Assessments
  Stenosis 0 - 25% | 50
  Stenosis >25 - 50% | 3
  Stenosis >50 - 75% | 1
  Stenosis >75% | 2
  Indeterminate | 8

8. Secondary Outcome: Number of Participants With Device-Related Adverse Events at 3 Years
Description: Number of participants with incidence of device-related adverse events at 3 year follow-up
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline
Number analyzed (Participants) | 107
Participants | 4

9. Secondary Outcome: Number of Participants With Device-related Adverse Events at 5 Years
Description: Subjects Observed with Device Related Adverse Events 5 years after Pipeline Placement
Time Frame: 5 years
Population: Subjects Observed with Device Related Adverse Events 5 years after Pipeline Placement
Measure: Count of Participants; unit: Participants
Arm/Group | Pipeline
Number analyzed (Participants) | 107
Participants | 2

ADVERSE EVENTS:
Time Frame: Cumulative incidence rate of adverse events observed at 5 years.
Arm/Group | Pipeline
Serious Adverse Events (participants affected / at risk) | 55/107
Other Adverse Events (participants affected / at risk) | 74/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pipeline (N=107)
Cerebral Haemorrhage (Nervous system disorders) | 6 (6)
Headcahe (Nervous system disorders) | 6 (6)
Cerebral Ischaemia (Nervous system disorders) | 3 (3)
Liird nerve disorder (Nervous system disorders) | 2 (2)
Ischaemia stroke (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Dimentia alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Vith nerve disorder (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Wolff-parkinson white syndrome (Cardiac disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 3 (3)
Ophthalmoplegia (Eye disorders) | 2 (2)
Retinal artery embolism (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intermittent claudification (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 3 (3)
Arterial aneurysm repair (Surgical and medical procedures) | 1 (1)
Intra-cerebral aneurysm repair (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Creast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Catheter site discharge (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disk degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pipeline (N=107)
Headache (Nervous system disorders) | 34 (34)
Visual Impairment (Eye disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 12 (12)
Infection (Infections and infestations) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6)
Paraesthesia (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No